CLINICAL TRIAL: NCT04368481
Title: Deep Learning for Identification of Abnormalities on Head MRI
Brief Title: MIDI (MR Imaging Abnormality Deep Learning Identification)
Acronym: MIDI
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: KCH18-197
Record Dates: First submitted 2020-02-18; First posted 2020-04-29 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Neurological Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study involves the development and testing of an artificial intelligence (AI) tool that can identify abnormalities using patient head scans conducted for routine clinical care and research volunteer scans. A deep learning algorithm will be developed using a dataset of retrospective and prospective MRI head scans to train, validate, and test convolutional networks using software developed at the Department of Biomedical Engineering, King's College London. The reference standard will be consultant radiologist reports of the MRI head scans.

DETAILED DESCRIPTION:
An automated strategy for identifying abnormalities in head scans could address the unmet clinical need for faster abnormality identification times, potentially allowing for early intervention to improve short- and long-term clinical outcomes. Radiologist shortages and increased demand for MRI scans lead to delays in reporting, particularly in the outpatient setting.

Furthermore, there is a wide variation in the management of incidental findings (IFs) discovered in 'healthy volunteers.' The routine reporting of 'healthy volunteer' scans by a radiologist poses logistical and financial challenges. It would be valuable to devise automated strategies to reliably and accurately identify IFs, potentially reducing the number of scans requiring routine radiological review by up to 90%, thus increasing the feasibility of implementing a routine reporting strategy.

Deep learning is a novel technique in computer science that automatically learns hierarchies of relevant features directly from the raw inputs (such as MRI or CT) using multi-layered neural networks. A deep learning algorithm will be trained on a large database of head MRI scans to recognize scans with abnormalities. This algorithm will be trained to classify a subset of these scans as normal or abnormal and then tested on an independent subset to determine its validity.

If the tested neural network demonstrates high diagnostic accuracy, future research participants and patients may benefit, as not all institutions currently review their research scans for incidental findings and clinical scans may not be reported for weeks in some cases. In both research and clinical scenarios, an algorithm could rapidly identify abnormal pathology and prioritize scans for reporting.

In summary, the aim is to develop a deep learning abnormality detection algorithm for use in both research and clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* All head MRI scans with compatible sequences
* > 18 years old

Exclusion Criteria:

* No corresponding radiologist report
* No consent for future use of the research images held within the historic database stored at The Centre for Neuroimaging Sciences (Kings College London).
* Poor image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult MRI head scan patients presenting at secondary and tertiary NHS centres across the UK for any indication.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of a convolutional neural network to recognise abnormalities on head MRI scans. | At end of study (5-year study)
  Sensitivity, specificity, positive predictive value, and negative predictive values.

SECONDARY OUTCOMES:
Sensitivity and specificity of a convolutional neural network to broadly categorise abnormalities on head MRI scans. | At end of study (5-year study)
  Sensitivity, specificity, positive predictive value, and negative predictive values.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Booth, Principal Investigator — King's College Hospital NHS Trust
Locations (33):
- United Kingdom (33):
  - Princess Royal University Hospital, King's College Hospital NHS Foundation Trust, Orpington, Kent
  - Buckinghamshire Healthcare Nhs Trust (Stoke Mandeville), Aylesbury
  - Mid and South Essex NHS Foundation Trust, Basildon
  - Bedfordshire Hospitals Nhs Foundation Trust, Bedford
  - Betsi Cadwaladr University Health Board, Bodelwyddan
  - East Kent Hospitals University Nhs Foundation Trust, Canterbury
  - South Eastern Health & Social Care Trust, Dundonald
  - Queen Victoria Hospital Nhs Foundation Trust, East Grinstead
  - Medway Nhs Foundation Trust, Gillingham
  - Northern Lincolnshire and Goole Nhs Foundation Trust, Grimsby
  - Calderdale and Huddersfield NHS Foundation Trust, Huddersfield
  - The Queen Elizabeth Hospital King'S Lynn Nhs Trust, Kings Lynn
  - Kingston Hospital Nhs Foundation Trust, Kingston
  - NHS FIFE, Kirkcaldy
  - Forth Valley Royal Hospital, Larbert
  - Leeds Teaching Hospital NHS Trust, Leeds
  - University Hospitals of Leicester Nhs Trust, Leicester
  - Kings' College Hospital, London
  - CNS, Maudsley Hospital, South London and Maudsley NHS Foundation Trust, London
  - Croydon University Hospital, Croydon Health Services NHS Trust, London
  - Guy's Hospital, Guy's and St Thomas's NHS Foundation Trust, London
  - St George's Hospital, St George's University Hospital NHS Foundation Trust, London
  - St Thomas' Hospital, Guy's and St Thomas's NHS Foundation Trust, London
  - Norfolk and Norwich University Hospitals Nhs Foundation Trust, Norwich
  - Queen's Medical Centre University Hospital, Nottingham University Hospitals NHS Foundation Trust, Nottingham
  - Surrey and Sussex Healthcare Nhs Trust, Redhill
  - East Sussex Healthcare Nhs Trust, Saint Leonards-on-Sea
  - Northern Lincolnshire and Goole Nhs Foundation Trust, Scunthorpe
  - Mid and South Essex Nhs Foundation Trust, Southend
  - St George'S University Hospitals Nhs Foundation Trust, Tooting
  - Torbay and South Devon Nhs Foundation Trust, Torquay
  - Royal Cornwall Hospitals Nhs Trust, Truro
  - West Hertfordshire Hospitals Nhs Trust, Watford

REFERENCES:
- [Derived] Wood DA, Guilhem E, Kafiabadi S, Al Busaidi A, Dissanayake K, Hammam A, Mansoor N, Townend M, Agarwal S, Wei Y, Mazumder A, Barker GJ, Sasieni P, Ourselin S, Cole JH, Nair N, Geetha A, Onyekwuluje C, Dineen R, Dhillon P, Costigan C, Fatania K, Igra M, Nichols R, Saada J, Juette A, Barbara RR, Spohr H, Booth TC; MIDI Consortium Group. Self-Supervised Text-Vision Alignment for Automated Brain MRI Abnormality Detection: A Multicenter Study (ALIGN Study). Radiol Artif Intell. 2026 Mar;8(2):e240619. doi: 10.1148/ryai.240619. PMID 41295086